CLINICAL TRIAL: NCT03890679
Title: Genomic Medicine for Ill Neonates and Infants (The GEMINI Study)
Acronym: GEMINI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); Children's Hospital Medical Center, Cincinnati (Other); MOUNT SINAI HOSPITAL (Other); University of North Carolina, Chapel Hill (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JHUSIRB00000007
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pediatric: Genetic Syndrome

STUDY DESIGN:
Intervention Model Description: Single Group - All participants underwent both rGS and NewbornDx.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients receiving genetic testing in the NICU (Experimental): The study included 400 probands, 388 mothers, and 316 fathers who participated
  Interventions: Diagnostic Test: rapid whole genomic sequencing (rWGS)

INTERVENTIONS:
Diagnostic Test: rapid whole genomic sequencing (rWGS) — rWGS and NewbornDx are genomic sequencing platforms
  Other Names: NewbornDx

SUMMARY:
The Genomic Medicine for Ill Neonates and Infants (The GEMINI Study) is a research study aimed at comparing the clinical and economic utility of performing rapid whole genomic sequencing versus a targeted genomic sequencing panel on neonates and infants suspected of having a genetic disorder. This study is funded by the National Institutes of Health.

This multicenter, prospective clinical trial will enroll 400 subjects at the Floating Hospital for Children at Tufts Medical Center (Boston, MA), Cincinnati Children's Hospital Medical Center (Cincinnati, OH), Mount Sinai Kravis Children's Hospital (New York, NY), North Carolina Children's Hospital (Chapel Hill, NC), Children's Hospital of Pittsburgh (Pittsburgh, PA), and Rady Children's Hospital (San Diego, CA).

DETAILED DESCRIPTION:
This multicenter, prospective clinical trial will examine the diagnostic yield and clinical utility of NewbornDx, a targeted genomic sequencing panel for use in the neonate, and rapid whole genomic sequencing (rWGS) testing in high-risk infants with signs/symptoms consistent with a possible genetic disorder. Infants will undergo NewbornDx and rWGS (proband) testing. The biological parent(s), when available, will undergo NewbornDx testing at the same time as the infant. For rWGS,the infant will undergo testing first. If a specific diagnosis that is consistent with the phenotype is not made with rWGS proband analysis alone, the parent(s) will undergo rWGS. The study will also evaluate the cost effectiveness of each test as well as standard of care (SOC) testing. A retrospective chart review of infants with suspected genetic disorders will be done to understand 1-year cost and health outcomes that would have been incurred in the absence of the advanced testing. The resulting data from the trial will be used in the economic evaluation comparing NewbornDx, rWGS, and SOC over a 1-year period and used as basis to simulate the lifetime cost-effectiveness of these testing strategies. A web-based clinical reference database to provide references, clinical management guidelines, opportunities for clinical trial participation, and support groups for each condition will be developed with separate interfaces for the parent/guardian(s) and medical provider. The clinical reference database will be qualitatively assessed by a survey of medical providers.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent from the parent/guardian
* Signs/symptoms consistent with a possible genetic disorder
* Admitted to a hospital participating in this study at the time of enrollment
* Less than one year corrected gestational age

Exclusion Criteria:

* A known genetic diagnosis (e.g. prenatal testing)
* Major congenital anomaly associated with a chromosomal anomaly detected on prenatal testing
* Presence of documented congenital infection
* Infants considered non-viable due to prematurity (< 23 0/7 weeks GA)

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill L Maron, MD, MPH, Principal Investigator — Women and Infants Hospital of Rhode Island; Jonathan M Davis, MD, Principal Investigator — Tufts Medical Center
Locations (6):
- United States (6):
  - Rady Children's Hospital - San Diego, San Diego, California
  - Tufts Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data that relates genomic data to phenotype or other biological states will be generated and released in accordance to the NIH GDS Policy. Data, including genome sequences (fastq files), variants (vcf files), and associated HIPAA compliant clinical metadata will be deposited in the Longitudinal Pediatric Data Resource (LPDR; https://www.nbstrn.org/research-tools/longitudinal-pediatric-data-resource). The LPDR, in turn, will deposit data in the NCBI dbGAP. Variants with ACMG recommended pathogenicity assessments will be deposited in ClinVar. Novel disorder gene assertions will be deposited in ClinGen (https://clinicalgenome.org/).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Annual data submissions supplemented by specific dataset deposits as manuscripts arising from this work are submitted for publication.
Access Criteria: Individual level data will be made available through controlled access. Genomic Summary Results will be made available through unrestricted access.

REFERENCES:
- [Result] Maron JL, Kingsmore S, Gelb BD, Vockley J, Wigby K, Bragg J, Stroustrup A, Poindexter B, Suhrie K, Kim JH, Diacovo T, Powell CM, Trembath A, Guidugli L, Ellsworth KA, Reed D, Kurfiss A, Breeze JL, Trinquart L, Davis JM. Rapid Whole-Genomic Sequencing and a Targeted Neonatal Gene Panel in Infants With a Suspected Genetic Disorder. JAMA. 2023 Jul 11;330(2):161-169. doi: 10.1001/jama.2023.9350. PMID 37432431
- [Result] Maron JL, Kingsmore SF, Wigby K, Chowdhury S, Dimmock D, Poindexter B, Suhrie K, Vockley J, Diacovo T, Gelb BD, Stroustrup A, Powell CM, Trembath A, Gallen M, Mullen TE, Tanpaiboon P, Reed D, Kurfiss A, Davis JM. Novel Variant Findings and Challenges Associated With the Clinical Integration of Genomic Testing: An Interim Report of the Genomic Medicine for Ill Neonates and Infants (GEMINI) Study. JAMA Pediatr. 2021 May 1;175(5):e205906. doi: 10.1001/jamapediatrics.2020.5906. Epub 2021 May 3. PMID 33587123
- [Derived] Lavelle TA, Maron JL, Kingsmore SF, Lin CH, Zhu Y, Sweigart B, Reed D, Gelb BD, Vockley J, Davis JM. Rapid Genome Sequencing Compared with a Gene Panel in Critically Ill Infants with a Suspected Genetic Disorder: An Economic Evaluation. J Pediatr. 2025 Nov 1;289:114889. doi: 10.1016/j.jpeds.2025.114889. Online ahead of print. PMID 41177396

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Genetic Testing for the Study: The study included 400 probands, 388 mothers, and 316 fathers who participated. They all received both rapid whole genomic sequencing (rWGS) and the NewbornDx panel which are genomic sequencing platforms
Period: Overall Study
Arm/Group | Patients Receiving Genetic Testing for the Study
Started | 400
Completed | 400
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Receiving Genetic Testing in the Study: The study included 400 probands, 388 mothers, and 316 fathers who participated
  rapid whole genomic sequencing (rWGS): rWGS and NewbornDx are genomic sequencing platforms
Arm/Group | Patients Receiving Genetic Testing in the Study
Number analyzed (Participants) | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 400
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 18 [8 to 66.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 114
  Not Hispanic or Latino | 286
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 7
  Black or African American | 43
  White | 208
  More than one race | 63
  Unknown or Not Reported | 53
Region of Enrollment [Number; unit: participants]
  United States | 400
Diagnostic yield [Number; unit: percentage] — The diagnostic yield for each group was calculated as percent that were positive for a pathogenic variant, likely pathogenic variant, or variant of uncertain significance (VUS). A VUS was only reported if it was present in a gene was located in or near a gene that was highly suspicious of causing the participant's phenotype.
  percentage | 49

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With a Confirmed Genetic Disorder Detected by NewbornDx
Description: If NewbornDx diagnoses a genetic disorder
Time Frame: 1-2 weeks
Population: Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Count of Participants; unit: Participants
Groups:
- the Number of Subjects With a Confirmed Genetic Disorder by Newborn Dx: 109 infants had a confirmed genetic disorder
Arm/Group | the Number of Subjects With a Confirmed Genetic Disorder by Newborn Dx
Number analyzed (Participants) | 400
Participants | 109

2. Primary Outcome: The Number of Subjects With a Confirmed Genetic Disorder Detected by rWGS
Description: If rWGS diagnoses a genetic disorder
Time Frame: 1-2 weeks
Population: Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Confirmed Genetic Disorder by rWGS: 195 patients received a diagnosis by rWGS alone
Arm/Group | Patients With a Confirmed Genetic Disorder by rWGS
Number analyzed (Participants) | 400
Participants | 195

3. Primary Outcome: Time in Hours to a Positive Result by NewbornDx
Description: Duration of time (hours) to determine diagnosis by NewbornDx
Time Frame: 1-2 weeks
Population: Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Time to Diagnosis by Newborn Dx: How many hours did it take to report out a result by Newborn Dx
Arm/Group | Time to Diagnosis by Newborn Dx
Number analyzed (Participants) | 400
hours | 100.3 [56.9 to 121.7]

4. Primary Outcome: Time in Hours to a Positive Result by rWGS
Description: Duration of time (hours) to determine diagnosis by rWGS
Time Frame: 1-2 weeks
Population: Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Time to Diagnosis by rWGS: How long did it take to report out results
Arm/Group | Time to Diagnosis by rWGS
Number analyzed (Participants) | 400
hours | 146.6 [79.3 to 237.8]

5. Primary Outcome: Perception of the Clinical Utility of Genomic Sequencing
Description: The Clinician Assessment of Clinical Utility assessed by physician survey using units on a likert scale with 1 meaning not useful at all and 5 meaning very useful. The Clinician Assessment of clinical utility was done collectively as a whole for both modes of genomic sequencing.
Time Frame: 1 week
Population: Physicians of record rated the overall utility of the genomic-sequencing process, based on collective results from both platforms using a 5-point Likert Scale (1, [not useful at all], to 5 [very useful]). Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Count of Participants; unit: Participants
Groups:
- Perception of Clinical Utility: Full analysis Cohort
Arm/Group | Perception of Clinical Utility
Number analyzed (Participants) | 398
Participants
  Very Useful | 150
  Useful | 152
  Neutral | 60
  Not very useful | 31
  Not useful at all | 5

6. Primary Outcome: Clinical Utility of Genomic Sequencing as Assessed by Changes in Clinical Care Management or Goals of Care
Description: The Clinician Assessment of Clinical Utility assessed by physician survey selecting the specific types of 35 possible management changes (i.e. surgical intervention implemented, medication changed, etc.) The intent was to examine any changes in care resulting from completing either genomic sequencing testing.
Time Frame: 1 week
Population: Changes were determined via follow-up with the physician of record (intensivist or geneticist). Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Count of Participants; unit: Participants
Groups:
- Changes in Management or Goals of Care: How many infants had changes in management or goals of care after the genetic testing was performed
Arm/Group | Changes in Management or Goals of Care
Number analyzed (Participants) | 400
Participants
  Any changes in care | 76
  Medication | 44
  Surgery | 23
  Withdrawal of life-sustaining support | 12
  Diet | 7
  Change in goal of care from comfort to cure | 3
  No changes in care | 235

7. Secondary Outcome: One Year Cost-effectiveness of Entire Cohort.
Description: Total cost of hospitalization, post-discharge follow-up until infant's 1 year CGA (corrected gestational age). Cost effectiveness of the cohort was measured across both sequence groups as a single group.
Time Frame: From enrollment to 1 year corrected gestational age
Population: A decision model simulated and compared total costs of rWGS from enrollment through 1 year corrected gestational age (study period) for: 1) early rGS, and 2) early NewbornDx followed by later rGS for undiagnosed infants. Model inputs included GEMINI data and 2023 Medicare rates; the primary outcome was total costs over the study period. Pre-specified in the protocol to assess and collect as a single group across both sequence tests.
Measure: Mean (Standard Deviation); unit: US dollars
Groups:
- Per Patient Cost Over a One-year Period With rWGS: Full cohort (infants with early testing and infants with late testing)
Arm/Group | Per Patient Cost Over a One-year Period With rWGS
Number analyzed (Participants) | 400
US dollars | 388,572 (31,271)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Full Cohort: Patients that underwent genetic testing with genomic sequencing and targeted neonatal gene sequencing test
Arm/Group | Full Cohort
All-Cause Mortality (participants affected / at risk) | 12/400
Serious Adverse Events (participants affected / at risk) | 0/400
Other Adverse Events (participants affected / at risk) | 12/400
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Cohort (N=400)
Genomic testing results reporting (Investigations) | 12 (12) — The reports were not sent encrypted to ensure confidentiality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03890679/Prot_SAP_001.pdf